CLINICAL TRIAL: NCT05462769
Title: Percutaneous Plug-based Arteriotomy Closure Device Use in Minimally Invasive Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Karolinska University Hospital
Other Study IDs: MANTA continued
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Minimally Invasive Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous vascular closure — Percutaneous arteriotomy closed using a plug-based arteriotomy closure device

SUMMARY:
A single-center prospective study. Patients undergoing minimally invasive cardiac surgery between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden are eligible. Femoral cannulation was performed percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA; Teleflex/Essential Medical, Malvern, PA). Data regarding preoperative clinical characteristics and operative details were obtained by medical records review.

ELIGIBILITY:
Inclusion Criteria:

* Operated with minimally invasive cardiac surgery between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden, with use of percutaneous femoral cannulation with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients operated with minimally invasive cardiac surgery between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden, with use of percutaneous femoral cannulation with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Any vascular groin-related complication | During the first 8 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma K, Kastengren M, Svenarud P, Green R, Dalen M. Routine use of percutaneous femoral cannulation in minimally invasive cardiac surgery. Eur J Cardiothorac Surg. 2023 Mar 1;63(3):ezad020. doi: 10.1093/ejcts/ezad020. PMID 36692172